CLINICAL TRIAL: NCT01684657
Title: A Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Tolerability of Asenapine With Flexible Dosing From 5mg to 20mg in Adults With Developmental Stuttering
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Study transferring to another facility
Sponsor: University of California, Irvine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Gerald Maguire, Senior Associate Dean, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Asenapine Stuttering
Record Dates: First submitted 2012-07-24; First posted 2012-09-13 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Stuttering
Keywords: Stuttering
MeSH Terms: conditions — Stuttering | interventions — asenapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): This is the comparator. Placebo will be matched to color, taste, size, and smell.
- Asenapine (Experimental): This is an atypical antipsychotic that blocks dopamine and increases serotonin. The dosage will be from 2.5 to 10mg daily throughout the study.
  Interventions: Drug: Asenapine

INTERVENTIONS:
Drug: Asenapine — This is an atypical antipsychotic that blocks dopamine and increase the serotonin level.
  Other Names: Saphris
  Arms: Asenapine

SUMMARY:
The purpose of this research study is to find out the potential benefits and safety of asenapine (Saphris®) in adults who suffer from the developmental form of stuttering.

It is hypothesized that individuals who are randomly assigned to asenapine will have an improvement in speech as compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

Subjects can be enrolled in the study only if they meet all of the following criteria:

1. Subjects must satisfy DSM-IV criteria for stuttering.
2. The nature of stuttering must be developmental in origin with the onset prior to ten years of age.
3. Subjects must have a score of moderate or higher on the SSI-IV. 4) Women of child-bearing potential are eligible to participate as long as they are practicing a medically accepted form of contraception (i.e. condom with spermicide or diaphragm, oral or depot contraception, or an intrauterine device).

5)Subjects will be male or female from the ages of 18-70. 6)Subjects will be of only English speaking.

Exclusion Criteria:

Subjects will be excluded from the study for any of the following reasons:

1. Stuttering related to a known neurologic cause (e.g. head trauma, stroke).
2. Unstable medical or psychiatric illness.
3. Active substance abuse within three months prior to study inclusion.
4. Any illness that would require the concomitant use of a CNS active medication during the course of the study.
5. Subjects with Parkinson's dementia or other degenerative neurologic illness.
6. Subjects who are pregnant or nursing an infant.
7. No minors (under the age of 18) will not be enrolled in this study as the research with this compound in children and adolescents has not been fully performed.
8. Subjects who suffer from seizures, irregular heartbeat or an elevated blood sugar level (glucose).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Stuttering Severity Instrument | 10 minutes
  This is an objective measure of stuttering in which it captures verbal samples of five minutes speaking during a conversation and 5 minutes of reading a passage.

SECONDARY OUTCOMES:
Clinical Global Impression | 2 minutes
  This is an evaluation of the patient by the investigator as to whether or not the subjects has improved, remained the same, or worsened while in the study.
Barnes Akathisia Scale | 3 minutes
  Measures how restless the subject is during the examination.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Maguire, M.D., Principal Investigator — UCIMC
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States